CLINICAL TRIAL: NCT07028931
Title: Effects of Visualization Technique Compared to Combined Stretching Protocol on Mindfulness and Performance in Racquet Sports
Brief Title: Effects of Visualization Technique Compared to Combined Stretching Protocol in Racquet Sports.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC 02059 ARINA ASAD
Record Dates: First submitted 2025-01-01; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Sport Injury
Keywords: visualization technique; mental imagery; combined stretching protocol; mindfulness; performance; racquet sports

STUDY DESIGN:
Intervention Model Description: Two groups will be formed. One group will be the visualization group, i.e., group A which will receive the mental imagery technique, which will take 15-20 minutes. Participants will be asked to start the session with breathing exercises, then move on to the visualization of the exercises, and then end the session with the visualization of the cool-down exercises. In Group A, participants will only visualize the protocol and will not perform it physically.
  In Group B, the participants will be asked to perform combined stretching protocol which will include warm-up, the protocol and then the cool-down exercises. This protocol will take 20 minutes.
  After performance readings will be taken in the 1st, 3rd and 6th weeks and data will be compared to find out which method is more effective to improve mindfulness and performance in racquet sports players.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visualization Technique (Experimental): This will include the visualization group, i.e., group A, which will receive the mental imagery technique, which will take 15-20 minutes. Participants will be asked to start the session with breathing exercises, then move on to the visualization of the exercises, and then end the session with the visualization of the cool-down exercises. In Group A, participants will only visualize the protocol and will not perform it physically.
  Interventions: Behavioral: Visualization technique
- Combined Stretching Technique (Active Comparator): In Group B, the participants will be asked to perform a combined stretching protocol, which will include a warm-up, the combined stretching protocol, i.e., hip flexor and hamstring combo, calf and Achilles stretch and spinal twist, and arm extension movements, and then the cool-down exercises, which will include hip flexor stretch, quadriceps stretch and calf stretch, biceps stretch, and triceps stretch. This protocol will take 20 minutes.
  Interventions: Other: Combined Stretching Protocol

INTERVENTIONS:
Behavioral: Visualization technique — In GROUP A, i.e., visualization technique Athletes will be shown a video of stretching protocols and then will be asked to visualize those exercises, the total session time will be approximately 20 minutes which will be divided into three phases: pre-Session visualization (5-10 minutes) which will begin with 1-2 minutes of deep breathing and mental preparation to start visualization technique then players will be asked to visualize dynamic stretching (leg swings, arm circles, and lunges) and static stretching (hamstring and shoulder stretch) for 2-3 minutes each. Then begins the during session visualization phase (1-2 minutes per stretch) the players will be asked to pause before each stretch to visualize the movements, muscle engagement and the feeling of stretch and the transit between the stretches and then last comes the post session phase of visualization (5 minutes) this will involve visualization of cool down exercises like spinal twist, bicep stretch, triceps and hip stretch.
  Arms: Visualization Technique
Other: Combined Stretching Protocol — GROUP B will receive Combined stretching training protocol. The overall duration will be 20 minutes starting from warm up (5-7 minutes) which will include light jogging arm swings, leg swings and lunges, hamstring and shoulder stretches then followed by combined stretching movements (8-10 minutes) this will include hip flexor and hamstring combo, calf and Achilles stretch and spinal twist and arm extension movements and ending with a cool down protocol (5-7 minutes) which will include hip flexor stretch, quadriceps stretch and calf stretch, bicep and triceps stretch.
  Arms: Combined Stretching Technique

SUMMARY:
This study intends to compare the effects of visualization technique with combined stretching protocol on racquet sports players to find out how these protocols affect their performance and mindfulness.

DETAILED DESCRIPTION:
In this study, two groups will be formed to find out the effects of visualization technique, i.e., mental imagery versus the combined stretching protocol, on racquet sports players over a course of 6 weeks. One group is given the mental imagery protocol, and the other group is given the combined stretching protocol, and at the end of the 1st, 3rd, and 6th weeks, readings are taken to compare the effects of these techniques on the mindfulness (awareness) and performance of the subjects enrolled in this study. A total of 52 participants will be involved, and the groups will be divided into 26, 26 each. Data will be analyzed through SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Males.
* Age 20 to 40 years.
* Not being able to concentrate/ focus well on the game.
* Amateur players with at least 1 year experience of playing Racquet sports.
* No current injuries or medical conditions that could affect participation in physical activities.
* Commitment to attend all training sessions and assessments

Exclusion Criteria:

* Players who are already familiar with visualization technique
* Recent chronic injuries that could impair performance or participation
* History of psychological disorder that might interfere with the training and assessment.
* Participation in other competitive sports that might confound the effects of intervention.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-02 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Mindfulness and Performance | 6 weeks approximately after the study starts
  This will assess the player's ability to stay focused and present in a moment during play and their performance, i.e., their ability to make decisions and their precision and accuracy in gameplay.

SECONDARY OUTCOMES:
Combined Stretching Protocol | 6 weeks approximately after the study starts
  the participants will be asked to perform combined stretching protocol which will include warm-up, the protocol and then the cool-down exercises. This protocol will take 20 minutes.
  After performance readings will be taken in the 1st, 3rd and 6th weeks and data will be compared to find out which method is more effective to improve mindfulness and performance in racquet sports players.

CONTACTS AND LOCATIONS:
Overall Officials: Riafat Mehmood, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No